CLINICAL TRIAL: NCT01639261
Title: Eine Phase II Studie über Interferon Gamma 1b Zur Behandlung Der steroidrefraktären Bronchiolitis Obliterans Nach Allogener SZT
Brief Title: A Phase II Trial on Treatment of Steroid-refractory Bronchiolitis Obliterans With Interferon Gamma 1b After Allogeneic SCT
Acronym: IFN_BOSZT_01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Regensburg (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Principal Investigator, Professor Ernst Holler MD, Senior physician, University Hospital Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFN_BOSZT_01; 2010-022467-36 (EudraCT Number)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Steroid-refractory Bronchiolitis Obliterans
Keywords: steroid-refractory; bronchiolitis obliterans; allogeneic stem cell transplantation; interferon gamma
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon gamma 1b — Initial dose: 50µg s.c. three times/week, without fever >38,5 dose increase: 50µg/m² BSA three times/week
  Other Names: Imukin

SUMMARY:
Improvement of quality of life in patients with BO and establishment of a new third line therapy

DETAILED DESCRIPTION:
Primary Objectives:

Objective improvement of lung function, i.e.:

* Improvement of SO2, pO2 or pCO2 in oxygen dependent or improvement of FiO2 in respiration dependent patients ≥ 20 % or
* Reduction of oxygen need in oxygen dependent patients ≥ 1L O2/min with constant parameters at blood gas analysis (BGA) or
* Improvement of obstructive parameters ≥ 20 % or
* Improvement of lung function score (LFS) at least about one grade Improvement of lung function should be detectable at least by two consecutive examinations of lung function or BGA within at least four weeks.

Secondary Objectives

* Morphological improvement of BO/BOOP at CT scan
* Reduction of steroids about at least 20 %

ELIGIBILITY:
Inclusion Criteria

* Allogeneic SCT
* Age ≥ 18 years
* BO, firmed by 2 out of 3 examinations:

  * Lung function/ BGA
  * CT scan in in- and expiration or
  * Histological diagnosis
* Therapy refractory BO, i.e. no improvement during at least three therapies, among:

  * Azithromycin + inhaled steroids/ bronchodilators
  * Systemic steroids 1 mg/kg BW
  * One of the following therapies: MMF, mTOR inhibitors or ECP
* Effective contraception (before, during and for 8 weeks after the treatment)
* Blood count: no severe neutropenia, defined as ANC > 1000/ml, platelets > 50/nl and haemoglobin > 8 g/dl
* Liver parameters (bilirubin, gammaGT, AP, ASAT, ALAT) lower than 3 x paramount normal range
* Kreatinin lower than 3 x paramount normal range
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Pregnant or nursing woman
* No appropriate contraception
* Participation in any other study within 4 weeks before or during the study
* Active acute GvHD of other organs than the lung > grade II or severe active chronic GvHD
* No appropriate antibiotic/ antimycotic therapy in documented infection
* Severe bone marrow suppression (ANC < 1000/ml) or graft failure
* Liver parameters (bilirubin, gammaGT, AP, ASAT and ALAT) higher than 3 x paramount normal range
* Kreatinin higher than 3 x paramount normal range
* Participation in another study within 4 weeks before or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
therapy response | 24 weeks
  Enhancement of therapy response from 15 % to 50 %

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Holler, Professor MD, Principal Investigator — University Hospital Regensburg
Locations (1):
- University Hospital Regensburg, Regensburg, Germany